CLINICAL TRIAL: NCT03821220
Title: Improving Physical Activity Levels in the Arabic- Speaking Residents of East Jerusalem With Prediabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Clalit Health Services (Other)
Collaborators: Hebrew University of Jerusalem (Other)
Responsible Party: Principal Investigator, Prof. Amnon Lahad, Director of Medical Quality unit and Chairman department of Family Medicine, Clalit Health Services, Jerusalem district, Clalit Health Services
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0201-17-COM2
Record Dates: First submitted 2019-01-24; First posted 2019-01-29 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Diabetes Mellitus
Keywords: Activity tracker; Arab population; Physical Activity
MeSH Terms: conditions — Diabetes Mellitus; Motor Activity | interventions — Fitness Trackers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Active Comparator): Patients will receive an activity tracker and written information for pre-diabetic, on top of their usual care.
  Interventions: Behavioral: Activity tracker plus usual care
- Group B (Active Comparator): Patients will receive an activity tracker, written information for pre-diabetic, and personalized physical activity prescription, on top of their usual care.
  Interventions: Behavioral: Activity tracker plus usual care; Behavioral: Personalized physical activity prescription
- Group C (Active Comparator): Patients will receive an activity tracker, written information for pre-diabetic, personalized physical activity prescription, three sessions of motivational interview support from trained physician assistants, and two session of dietitian support, on top of their usual care.
  Interventions: Behavioral: Motivational Interview support and Dietitian support; Behavioral: Activity tracker plus usual care; Behavioral: Personalized physical activity prescription

INTERVENTIONS:
Behavioral: Motivational Interview support and Dietitian support — Three sessions of a structured motivational support intervention. Each patient will be required to set a SMART physical activity personal objective. The sessions will cover possible barriers and facilitators, enhancing self-efficacy, and feedback. In addition two sessions with a dietitian to discuss ways to improve current health habits.
  Arms: Group C
Behavioral: Activity tracker plus usual care — Each patient will receive their own activity tracker (vivofit 3) with instructions on use, in addition to usual care, and written handouts for pre-diabetic patients.
Behavioral: Personalized physical activity prescription — Each patient will receive a personalized prescription of recommended physical activity including type of activity, duration and frequency.
  Arms: Group B; Group C

SUMMARY:
This three-arm clinical trial aims to improve levels of physical activity among Arabic- speaking residents of East Jerusalem with prediabetes. Levels of daily physical activity (assessed through activity trackers), dietary habits and self-assessed health will be compared between patients that receive only the activity tracker and written information (group A), receive the activity tracker, written information and a personalized physical activity prescription (group B), and those that receive in addition also intensive follow-up with motivational interview by physician assistants and a dietitian (group C)

DETAILED DESCRIPTION:
This is a three-arm clinical trial studying the effect of providing activity trackers with intensive motivational interview by trained physician assistants, and dietitian counselling, on the levels of daily physical activity among Arabic- speaking residents of East Jerusalem with prediabetes from Clalit Health Services. In addition, this study will also assess healthy dietary changes, and self assessed health and quality of life.

The study will compare three groups (total 375, each group 125):

Group A - will receive activity trackers and written educational handouts in addition to their usual care.

Group B - will receive all of group A intervention components and also a personalized physical activity prescription.

Group C - will receive all of group B components and also intensive motivational interview support by trained physician assistants (3 sessions), and dietitian support (two sessions).

Each participant will be followed-up for six months, with data collection occurring at baseline, three months and six months. Data collection will include average weekly steps, blood pressure, anthropometric measurements, routine blood tests (including fasting glucose, HbA1C, and lipid profile), physical activity survey, Mediterranean dietary habits survey, Food Frequency Questionnaire, and quality of life survey.

ELIGIBILITY:
Inclusion Criteria:

Pre-diabetes patients - Impaired fasting glucose at least twice between 100-125 mg/dL in the two years prior to the study; or HbA1C 5.7%-6.4% twice in the two years prior to the study; or one test of fasting glucose of 100-125 mg/dL, and one test of HbA1C between 5.7%-6.4% in the two years prior to the study.

Exclusion Criteria:

1. Diabetes including a doctor's diagnosis based on a medical file or a recurrence of fasting blood glucose values above 126 mg/dL in the year preceding the study or a glucose value greater than 200 mg/dL in the year prior to the study or HbA1C above 6.5%
2. Treatment with diabetes drugs other than metformin, as prescribed in the medical file with regular or chronic medications
3. Artificial lower limbs or inability to walk normally (eg: stroke with plegia)
4. Chronic obstructive pulmonary disease
5. Known heart disease (with impaired exercise tolerance)
6. Pregnancy
7. Medical conditions:

   * a cardiac event/ Transient ischemic attack in the last year
   * Cerebrovascular attack with residual impairment
   * Surgery that required hospitalization in the last year
   * Injury to lower limbs that prevents regular walking
   * Malignancy excluding skin cancer small cell carcinoma or basal cell carcinoma

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Estimated)
Dates: Start 2019-02-15 (Estimated); Primary Completion 2021-02-15 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Physical activity level assessed through average weekly steps | six months

SECONDARY OUTCOMES:
Fasting glucose levels | six months
HbA1C levels | six months
Body Mass Index | six months
Lipid profile | six months
Blood pressure | six months
Energy intake 500< kcal/d <6000 kcal/d | Six months
Waist circumference | six months
Fat intake 15 <gram/day<200 | six months
Protein intake 10<gram/day<300 | six months
Iron intake 0<mg/day<50 | six months
Folic acid intake 15< μg/day<3000 | six months
Vitamin A intake 20< μg RAE/day<2500 | six months
Vitamin C intake 0<mg/day<2500 | six months

CONTACTS AND LOCATIONS:
Overall Officials: Amnon Lahad, MD, Principal Investigator — Clalit

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared